CLINICAL TRIAL: NCT03063996
Title: Peripheral Internal Jugular Vein ('Peripheral IJ') Access in Patients Identified as Difficult Intravenous Access Research Study
Brief Title: Peripheral Internal Jugular Vein ('Peripheral IJ') Access in Patients Identified as Difficult Intravenous Access
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: A16-598
Record Dates: First submitted 2017-02-16; First posted 2017-02-24 (Actual); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Difficult IV Access

STUDY DESIGN:
Intervention Model Description: This will be a randomized control trial comparing peripheral IJ to standard care of difficult access patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (peripheral IV access) (Other): Patient with a history of difficult access or a patient that currently has difficult peripheral IV access.
  Interventions: Procedure: peripheral IV access procedure
- Peripheral IJ access (Active Comparator): Patient with a history of difficult access or a patient that currently has difficult peripheral IV access and is randomized into the group that gets peripheral IJ access.
  Interventions: Procedure: Peripheral IJ access procedure

INTERVENTIONS:
Procedure: peripheral IV access procedure — standard of care guided IV access into peripheral vein excluding IJ
  Arms: Standard of Care (peripheral IV access)
Procedure: Peripheral IJ access procedure — standard of care guided IV access into IJ
  Arms: Peripheral IJ access

SUMMARY:
The primary aim of this study is to determine if the insertion of a peripheral Internal Jugular (IJ) catheter is faster than a standard of care intravenous (IV)access in patients with difficult access. The secondary aims of this study examine patient discomfort between standard IV insertion vs. peripheral IV insertion as well as a comparison of complication rates between the two methods of insertion. Support for the peripheral IV procedure could provide an option for the thousands of Emergency Department (ED) patients who daily encounter the situation of difficult IV access and the numerous needle pokes that accompany it. Using this procedure may result in greater patient satisfaction and reduced complication rates.

DETAILED DESCRIPTION:
This will be a randomized control trial comparing peripheral IJ to standard care of difficult access patients.

1. Patients will be identified by nurses as having difficult IV access. This can be determined based on past history or immediate experience. In other words, while a nurse is caring for a patient, s/he might notice that the patient looks to have difficult veins for an IV and may ask the patient 'Are you a hard stick?'. On the other hand, the nurse may fail at a number of attempts at placing an IV. In both of the cases, the patients can be determined to have difficult access and the nurse will have the option to contact the research assistant or continue with current attempts.
2. Nurse will contact research assistant.
3. Research assistant (RA) will determine if the patient is being cared for by an MD with appropriate experience for placing the peripheral IJ (attending, second or third year ED resident).
4. RA will consent patient, discussing possible continuation of IV or IJ catheter insertion. If patient agrees, he/she will be enrolled in the study.
5. Patient will be randomized.
6. Time clock will be started by RA when nurse or study member (attending physician, second or third year resident) start the procedure (IV or IJ).
7. RA will monitor procedure progress and stop time clock when access has been confirmed by study member or by nurse.
8. RA will survey patient regarding pain during procedure and satisfaction.
9. Patient chart will be queried at the completion of ED visit or hospitalization for complications. Chart will be queried again at two weeks to evaluate for any return visit complication.

Catheters will be placed by attending physicians and residents (2nd and 3rd years) with experience placing ultrasound guided internal jugular central venous catheters. Because the procedure is identical to the first step of placing an IJ Central Venous Catheter, there is no special training needed for the procedure itself. A video will be created and viewed by all placing the catheters to show the specifics so that there is standardization between individuals.

Attempts to place the peripheral IJ will be limited to two. If not successful after two attempts, the patient will return to 'standard care' and the treatment team will decide on further directions such as ultrasound guided peripheral IV or central venous line.

ELIGIBILITY:
Inclusion Criteria:

1. Emergency Department patient
2. Need for IV access
3. Difficult access as determined by nurse based on current challenges with IV access or in discussion with patient regarding past experience
4. Patient in stable condition as determined by treating team
5. English speaking
6. Ability to consent
7. Age ≥ 18 years

Exclusion Criteria:

1. Prior neck surgery
2. Known blood clot in IJ vein
3. Overlying infection
4. Need for immediate IV access
5. Provider not available for procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-02-07 (Actual); Primary Completion 2018-06-05 (Actual); Study Completion 2018-06-12 (Actual)

PRIMARY OUTCOMES:
Total time to gain successful IV access | ED arrival to successful venous access, up to 300 minutes
  Time to successful IV (or IJ) access in minutes from ED arrival

SECONDARY OUTCOMES:
Venous access complication | Up to 2 weeks after IV placement and/or removal
  Variables: Immediate Complications -noted at time of procedure (hematoma, arterial puncture, pneumothorax, infection, line failure) Delayed complications - noted at time of discharge OR at 2 week chart follow-up (hematoma, pneumothorax, infection, line failure)
Procedural patient comfort | Average 5 minutes to 1 hour post procedure
  Pain-score assessment (10-point Likert scale)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Zwank, MD, Principal Investigator — Regions Hospital
Locations (1):
- Regions Hospital, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to share individual personnel data